CLINICAL TRIAL: NCT06293274
Title: The Effect of Discharge Education on Maternity Blues and Postpartum Depression
Brief Title: The Importance of Discharge Education for Mommy Blues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, sena dilek, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: sdilek5
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Postpartum Sadness
Keywords: discharge; maternity; sadness; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discharge education (Experimental): Participants assigned to the discharge education group will receive discharge education about postpartum blues and postpartum depression. A "Personal Information Form" will be used. Discharge training and data collection are expected to take approximately 15-20 minutes. 5-7 days postpartum after the mothers are discharged. The 32-item "Motherhood Sadness Scale" will be administered by the researcher by telephone during the following days. In the 6th week of the postpartum period, the mothers will be contacted by the researcher by telephone and the 10-item "Edinburgh Postpartum Depression Scale" will be administered.
  Interventions: Procedure: Discharge training
- Routine discharge training (No Intervention): Participants assigned to the routine discharge training group will receive routine discharge training. "A personal information form will be used. Discharge training and data collection are expected to take approximately 15-20 minutes. 5-7 days postpartum after mothers are discharged. The 32-item "Motherhood Sadness Scale" will be administered by the researcher by telephone during the following days. In the 6th week of the postpartum period, the mothers will be contacted by the researcher by telephone and the 10-item "Edinburgh Postpartum Depression Scale" will be administered.

INTERVENTIONS:
Procedure: Discharge training — What is motherhood blues? Why does it occur? What are its symptoms? How to deal with it? What is postpartum depression? What causes postpartum depression? Information is provided on this topic.
  Other Names: motherhood blues education
  Arms: Discharge education

SUMMARY:
The study will be conducted with participants who will give birth at Farabi Training and Research Hospital in Darıca District, Kocaeli Province.

The sample size of the study was calculated using the G*Power 3.1.9.2 program, and the effect size of the Edinburgh Postnatal Depression Scale (EPDS) score in the Sun et al. (2021) study was considered in the effect size calculation. In the relevant article, the effect size is reported as effect size: 0.47. In our planned research, the minimum number of individuals to be sampled was calculated using G*Power 3.1.9.2 with effect size: 0.47 α= 0.05, power: 0.80, and the sample size was set at a minimum of 57 participants in each group. In anticipation of possible data loss, the study will be completed with a total of 140 participants, including 70 cases and 70 routine discharge training groups. This research aims to determine the effect of discharge training on maternal blues and postpartum depression on the levels of maternal blues and postpartum depression during postpartum follow-up.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of discharge training on maternal sadness and postpartum depression on the level of maternal sadness and postpartum depression in the puerperium follow-up. In this context, the hypotheses of the study are as follows;

Hypothesis 1:

H0: There is no difference in the total scores of the Maternal Sadness Scale used in the postpartum follow-up of mothers who received discharge training on maternal sadness and postpartum depression and mothers who did not receive training.

H1: There will be a difference in the total scores of the Maternal Sadness Scale used in the postpartum follow-up of mothers who received discharge education on maternal sadness and postpartum depression and mothers who did not receive education.

Hypothesis 2:

H0: There will be no difference in total scores on the Edinburgh Postpartum Depression Scale used in the postpartum follow-up of mothers who received discharge education on maternal grief and postpartum depression and mothers who did not receive education.

H1: There is a difference in the total scores of the Edinburgh Postpartum Depression Scale used in the postpartum follow-up of mothers who received discharge education on maternal grief and postpartum depression and mothers who did not receive education.

Mothers enrolled in the study will be randomly assigned to groups, and homogeneity in the distribution of groups will be ensured. "Random Allocation Software Program will be used to randomly assign mothers to groups, and a randomization list for the study will be generated by determining the number and group number of each participant.

Postpartum women to be included in the study will be assigned to one of the routine discharge training and discharge education groups by the researcher according to the order in the randomization list. Only that mother will be studied until the mother assigned to the randomization group has been informed about the research and has completed the necessary training compared to the routine discharge training/discharge education group. After the mother's research process is completed, another mother who has been admitted to the ward and meets the research criteria will be assigned to the other group on the randomization list and the necessary practices will be carried out. If the mother leaves the study for any reason during the study, the first mother admitted to the ward who meets the research criteria will be assigned to the other group on the randomization list.

In a randomized controlled trial with discharge education and routine discharge training groups, after the research groups are formed; In the first phase, the participants assigned to the discharge education group will be given a discharge education on postpartum depression and motherhood blues through a face-to-face interview technique and a "personal information form" will be used. It is expected that the discharge training and data collection will take approximately 15-20 minutes. After the training, an information booklet prepared by the researchers after a literature review will be given to the participants in print, via email or WhatsApp, depending on the researcher's preference. 5-7 days of postpartum period after the mothers are discharged. On these days, the researcher will call you and inform you that the 32-item Motherhood Sadness Scale will be administered. Data collection is expected to take approximately 5-10 minutes. Interviewed mothers will be contacted by the researcher by telephone at 6 weeks postpartum after discharge from the hospital and informed that the 10-item Edinburgh Postpartum Depression Scale will be administered. Data collection is expected to take approximately 5 minutes.

After the scale data are collected during the interview, the researcher will provide brief verbal information about the Motherhood Blues Scale and the Edinburgh Postpartum Depression Scale scores, and mothers whose scale scores are determined to be high will be referred to the necessary units to increase necessary psychiatric counseling and social support.

The mother assigned to the routine discharge training group will receive routine hospital discharge education. Then the "Personal Information Form" will be used. The mother whose contact information was collected will be examined by the researcher on the 5th-7th day of her postpartum period after her discharge. On these days, the researcher will call you and inform you that the 32-item "Motherhood Sadness Scale" will be administered. Data collection is expected to take approximately 5-10 minutes. Interviewed mothers will be contacted by the researcher by telephone at 6 weeks postpartum after discharge from the hospital and informed that the 10-item Edinburgh Postpartum Depression Scale will be administered. Data collection is expected to take approximately 5 minutes. After the scale data have been collected during the interview, the researcher will provide brief verbal information about the Motherhood Blues Scale and Edinburgh Postpartum Depression Scale scores, and mothers whose scale scores are determined to be high will be referred to the necessary services to enhance necessary psychiatric care and social support.

ELIGIBILITY:
Inclusion Criteria:

* 38-42. Those who gave birth between weeks of gestation,
* Those who have had vaginal birth or caesarean section,
* Able to speak and understand Turkish,
* Those over 18 years of age,
* Mothers with a single healthy baby
* Those with an Edinburgh Postnatal Depression Scale score of 9 or less in depressive symptoms screening

Exclusion Criteria:

* Preterm or postterm birth,
* Received psychiatric treatment or used psychotropic medications during pregnancy,
* Having a history of substance dependence and/or use in the past 6 months,
* Being in the high-risk category,
* Interventional/instrumented birth (Kiwi, vacuum, crystal maneuver),
* Mothers having babies with congenital malformations requiring intensive care intervention (small for gestational age, mort de fetus, fetus without major pathology according to ultrasonography).
* Participants who wish to withdraw from the study at any time will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 140 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Motherhood Sadness Scale | 5-7 days of the postpartum period after the mother's discharge. It will be obtained by the researcher by telephone on the following days.
  The scale developed to evaluate motherhood blues consists of 32 items and 8 sub-dimensions. These sub-dimensions; skin-to-skin contact, communication, staying in the same room, breastfeeding, physical adaptation, responsibility, culture, economic factors, information and economic support, social support. Scale items contain positive and negative expressions. The scale is graded as 'completely appropriate (5 points), appropriate (4 points), rarely appropriate (3 points), not appropriate (2 points), not at all appropriate (1 point). The minimum score that can be obtained from the scale is 32 and the maximum score is 160. A high total score in the evaluation of the scale indicates experiencing motherhood blues.
Edinburgh Postnatal Depression Scale - EPDS | At 6 weeks postpartum, the researcher will call and administer the 10-item Edinburg Postpartum Depression Scale.
  The scale consists of 10 items. Items are evaluated in a 4-point Likert format and scored between 0-3. The lowest score that can be obtained from the scale is 0 and the highest score is 30. Although the cut-off scores for the scale vary between studies, it is stated that a cut-off score of 12 may be sufficient to determine clinical depression. The scale is a screening scale to determine the risk of postpartum depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sena Dilek Aksoy, Ph.D., Study Director — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Background] Sun Y, Li Y, Wang J, Chen Q, Bazzano AN, Cao F. Effectiveness of Smartphone-Based Mindfulness Training on Maternal Perinatal Depression: Randomized Controlled Trial. J Med Internet Res. 2021 Jan 27;23(1):e23410. doi: 10.2196/23410. PMID 33502326